CLINICAL TRIAL: NCT00356551
Title: Family Strengthening in Native Communities Project
Brief Title: Family Spirit Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency); Annie E. Casey Foundation (Other Government); Ford Foundation (Other); Charles Stewart Mott Foundation (Other); Educational Foundation of America (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1 UDI SPO9588
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Substance Abuse
Keywords: Teen pregnancy; Family strengthening; Substance abuse prevention; Depression prevention; Parent involvement
MeSH Terms: conditions — Substance-Related Disorders

INTERVENTIONS:
Behavioral: Family Spirit curriculum

SUMMARY:
The goals of this study are to evaluate the effects of an in-home parenting education program, called Family Spirit, on parenting knowledge and skills and decreasing alcohol and substance use compared to a breast-feeding education. In addition, we will assess aspects of mother/child interaction.

DETAILED DESCRIPTION:
To evaluate the study, we employed a randomized controlled design using a blocked randomization procedure. In this procedure, single woman and women with a participating father were randomized in equal numbers to the Family Spirit or the breast-feeding education program.

Both treatment and comparison groups were assessed at multiple times. The number of times depended on when the participant was recruited into the program. Women recruited into the program between the study's start (May 2002) and January 31, 2004 were assessed at four times: 1) The Pre-test occurs after informed consent (occurring at least 16 weeks before the birth of the infant), 2) The Mid-Test at 6-8 weeks after the delivery of the infant, 3) The Post-Test at 6 months post-partum (which is the end of the intervention period), and 4) The 6-month Follow Up Test occurs at 1 year post-partum. Women recruited into the program between February 1, 2004 and March 31, 2004 (the date recruitment ended) were assessed at three times: 1) The Pre-test occurs after informed consent (occurring at least 16 weeks before the birth of the infant), 2) The Mid-Test at 6-8 weeks after the delivery of the infant, and 3) The Post-Test at 6 months post-partum (the end of the intervention period).

Family Health Educator (FHE)s also conducted two instruments specific to child development: the HOME and the ITSEA. The Home Observation for Measurement of the Environment (HOME) was administered at the Post-Test and Follow-Up points (just the post-point for women recruited into the study between February 1, 2004 and March 31, 2004). This measure was an observatory measure completed by FHEs and provided a systematic measurement of the family environment. The Infant-Toddler Social and Emotional Assessment (ITSEA) was a self-report form completed by parents at their Follow-Up visit (not completed for women recruited into the study between February 1 and March 31, 2004). This measure assessed social-emotional problems and competencies in 12- to 36-month olds. FHEs also administered a Client Satisfaction Scale to mothers in the (Family Support Person) FSP group who completed their participation in the program. This Scale assessed their satisfaction with the various curricular sections and their FHE.

ELIGIBILITY:
Inclusion Criteria:

* Native American pregnant teens or young women ages 12-22 years old at the time of conception.
* Women ages 20-22 years at the time of conception must be pregnant for the first time.
* Partners of pregnant teens must be between the ages of 12-24.
* Pregnant <28 weeks gestation and able to meet the requirements for completing the program in a timely way.
* An enrolled tribal member.
* Reside in the Reservation Service Unit Catchment Area and within 60 mile of the Indian Health Service Unit Headquarters.

Exclusion Criteria:

* Severe mental illness - schizophrenia, bipolar disorder, incapacitating depression, or Substance abuse/dependence in need of intensive and specific treatment
* Active legal problems - subjects will not be enrolled if they are incarcerated or if program participation has been made a condition of parole
* Ongoing social service involvement for abuse and neglect

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 320
Dates: Start 2002-05; Study Completion 2005-09

PRIMARY OUTCOMES:
Increase in parent knowledge, measured at baseline, 2 weeks post-partum, 6 months post-partum and 12 months post-partum
Increase in parent skills, measured at baseline, 2 weeks post-partum, 6 months post-partum and 12 months post-partum
Decrease in parental high-risk behaviors, measured at baseline, 2 weeks post-partum, 6 months post-partum and 12 months post-partum
Increase in parental-child involvement, measured at baseline, 2 weeks post-partum, 6 months post-partum and 12 months post-partum

CONTACTS AND LOCATIONS:
Overall Officials: John Walkup, MD, Principal Investigator — Johns Hopkins University; Allison Barlow, MA, MPH, Study Director — Johns Hopkins Center for American Indian Health
Locations (5):
- United States (5):
  - Johns Hopkins Center for American Indian Health, Fort Defiance, Arizona
  - Johns Hopkins Center for American Indian Health, Tuba City, Arizona
  - Johns Hopkins Center for American Indian Health, Whiteriver, Arizona
  - Johns Hopkins Center for American Indian Health, Baltimore, Maryland
  - Johns Hopkins Center for American Indian Health, Gallup, New Mexico

REFERENCES:
- [Derived] Walkup JT, Barlow A, Mullany BC, Pan W, Goklish N, Hasting R, Cowboy B, Fields P, Baker EV, Speakman K, Ginsburg G, Reid R. Randomized controlled trial of a paraprofessional-delivered in-home intervention for young reservation-based American Indian mothers. J Am Acad Child Adolesc Psychiatry. 2009 Jun;48(6):591-601. doi: 10.1097/CHI.0b013e3181a0ab86. PMID 19454915